CLINICAL TRIAL: NCT05092360
Title: A Phase 3, Multicenter, Open-Label, Randomized Study of Nemvaleukin Alfa in Combination With Pembrolizumab Versus Investigator's Choice Chemotherapy in Patients With Platinum-Resistant Epithelial Ovarian, Fallopian Tube, or Primary Peritoneal Cancer (ARTISTRY-7)
Brief Title: Phase 3 Study of Nemvaleukin Alfa in Combination With Pembrolizumab in Patients With Platinum-Resistant Epithelial Ovarian Cancer (ARTISTRY-7)
Acronym: ARTISTRY-7
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study terminated due to business and strategic decision.
Sponsor: Mural Oncology, Inc (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ALKS 4230-007; GOG-3063 (Other: The GOG Foundation); ENGOT-OV68 (Other: European Network Gynaecological Oncological Trial groups); KEYNOTE-C71 (Other: Merck); APGOT-OV8 (Other: APAC Gynecologic Oncology Trial Group)
Record Dates: First submitted 2021-10-13; First posted 2021-10-25 (Actual); Results first posted 2025-08-28 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-06

CONDITIONS: Platinum-resistant Ovarian Cancer; Fallopian Tube Cancer; Primary Peritoneal Cancer
Keywords: PROC; EOC; ALKS 4230; IL-2; Ovarian Cancer; KEYNOTE-C71; Platinum Resistant; Epithelian Ovarian Cancer; Nemvaleukin alfa; Pembrolizumab; ARTISTRY-7; ART-7; paclitaxel; pegylated liposoma doxorubicin; PLD; topotecan; gemzar; gemcitabine
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms | interventions — pembrolizumab; liposomal doxorubicin; Doxorubicin; Paclitaxel; Taxes; Topotecan; Gemcitabine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Nemvaleukin and Pembrolizumab Combination (Experimental)
  Interventions: Biological: Nemvaleukin and Pembrolizumab Combination
- Pembrolizumab (enrollment completed) (Experimental)
  Interventions: Biological: Pembrolizumab
- Nemvaleukin (enrollment completed) (Experimental)
  Interventions: Biological: Nemvaleukin
- Investigator's Choice (Active Comparator): Options for protocol-specific Investigator's choice chemotherapy include one of the following: pegylated liposomal doxorubicin (PLD), paclitaxel, topotecan, or gemcitabine. The Investigator will pre-select the Investigator's choice treatment before the randomization of each patient.
  Interventions: Drug: Pegylated Liposomal Doxorubicin (PLD); Drug: Paclitaxel; Drug: Topotecan; Drug: Gemcitabine

INTERVENTIONS:
Biological: Nemvaleukin and Pembrolizumab Combination — Nemvaleukin: 6 µg/kg/day; Days 1 through 5 of 21-day cycles; IV infusion over 30 minutes and Pembrolizumab: 200 mg; Day 1 of 21-day cycles; IV infusion over 30 minutes
  Other Names: Nemvaleukin alfa; ALKS 4230; Keytruda
  Arms: Nemvaleukin and Pembrolizumab Combination
Biological: Pembrolizumab — Pembrolizumab: 200 mg; Day 1 of 21-day cycles; IV infusion over 30 minutes
  Other Names: Keytruda
  Arms: Pembrolizumab (enrollment completed)
Biological: Nemvaleukin — Nemvaleukin: 6 µg/kg/day; Days 1 through 5 of 21-day cycles; IV infusion over 30 minutes
  Other Names: Nemvaleukin alfa; ALKS 4230
  Arms: Nemvaleukin (enrollment completed)
Drug: Pegylated Liposomal Doxorubicin (PLD) — 40 mg/m2; Day 1 of 28-day cycles; IV infusion; 1 mg/min (Cycle 1); 60 min infusion (Cycles 2+)
  Other Names: PLD- CAELYX; DOXIL; LIPODOX; Myocet
  Arms: Investigator's Choice
Drug: Paclitaxel — 80 mg/m2; Days 1, 8, 15, and 22 of 28-day cycles; IV infusion over 60 min
  Other Names: Nov-Onxol; Taxol; Onxol; Paclitaxel Novaplus
  Arms: Investigator's Choice
Drug: Topotecan — 4 mg/m2; Days 1, 8, and 15 of 28-day cycles; or 1.25 mg/m2, Days 1 through 5 of 21-day cycles; IV infusion over 30 min
  Other Names: Hycamtin; Potactasol
  Arms: Investigator's Choice
Drug: Gemcitabine — 1,000 mg/m2; Days 1 and 8 of 21-day cycles; IV infusion over 30 min
  Other Names: Gemzar; Infugem
  Arms: Investigator's Choice

SUMMARY:
This is a Phase 3, multicenter, open-label, randomized study of nemvaleukin in combination with pembrolizumab versus protocol-specific Investigator's choice chemotherapy in patients with platinum-resistant epithelial ovarian, fallopian tube, or primary peritoneal cancer.

DETAILED DESCRIPTION:
Patients will be centrally allocated in a randomized fashion (3:1:1:3) to receive either:

Arm 1: Nemvaleukin and pembrolizumab combination therapy Arm 2: Pembrolizumab monotherapy Arm 3: Nemvaleukin monotherapy Arm 4: Investigator's choice chemotherapy include one of the following: pegylated liposomal doxorubicin (PLD), paclitaxel, topotecan, or gemcitabine.

ELIGIBILITY:
Inclusion Criteria:

* Patient is female and ≥18 years of age.
* Patient has histologically confirmed diagnosis of EOC (ie, high-grade serous, endometrioid of any grade, clear cell), fallopian tube cancer, or primary peritoneal cancer.
* Patient has platinum-resistant/refractory disease, defined as disease progression within 180 days following the last administered dose of platinum therapy beyond first-line setting (resistant) or lack of response or disease progression while receiving the most recent platinum-based therapy (refractory). Patient must have progressed radiographically on or after their most recent line of anticancer therapy.
* Patient must have received at least 1 prior line of systemic anticancer therapy in the platinum sensitive setting, and no more than 5 prior lines of systemic anticancer therapy in the platinum-resistant setting. Patient must have received at least 1 line of therapy containing bevacizumab.
* Patient has at least one measurable lesion that qualifies as a target lesion based on RECISTv1.1.
* Patient is willing to undergo a pre-treatment tumor biopsy or provide qualifying archival tumor tissue.

Exclusion Criteria:

* Patient has primary platinum-refractory disease or primary platinum resistance, defined as disease progression during first-line platinum-based therapy (refractory) or disease progression <3 months after completion of first-line platinum-based therapy (resistant).
* Patient has histologically confirmed diagnosis of EOC with mucinous or carcinosarcoma subtype.
* Patient has nonepithelial tumor (eg, germline or stromal cell tumor) or ovarian tumor with low malignant potential (ie, borderline or low-grade serous tumor).
* Patient requires fluid drainage (eg, paracentesis, thoracentesis, pericardiocentesis) of ≥500 mL within 4 weeks of first dose of study drug.
* Patient has received prior IL-2-based or IL-15-based cytokine therapy; patient has had exposure, including intralesional, to IL-12 or analogs thereof.
* Patient has prior exposure to any anti-PD1/PD-L1 therapy.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 456 (Actual)
Dates: Start 2022-01-10 (Actual); Primary Completion 2025-01-08 (Actual); Study Completion 2025-05-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mural Oncology Medical Monitor, Study Director — Mural Oncology, Inc
Locations (117):
- United States (37):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Alaska Women's Cancer Care, Anchorage, Alaska
  - Arizona Oncology, Tucson, Arizona
  - University of California, San Diego (UCSD)- Moores Cancer Center, La Jolla, California
  - University of California, Los Angeles (UCLA), Los Angeles, California
  - Ventura County Hematology- Oncology, Oxnard, California
  - University of Florida (UF) Health Cancer Center - Orlando Health, Orlando, Florida
  - Sarasota Memorial Hospital, Sarasota, Florida
  - Emory University, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - Indiana University (IU), Indianapolis, Indiana
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - University of Maryland School of Medicine, Baltimore, Maryland
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Trinity Health Ann Arbor Hospital, Ypsilanti, Michigan
  - Astera Cancer Care, East Brunswick, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - University of New Mexico, Albuquerque, New Mexico
  - Womens Cancer Care Associates, Albany, New York
  - Westchester Medical Center, Hawthorne, New York
  - NYU Langone Health, New York, New York
  - David H. Koch Center for Cancer Care at Memorial Sloan Kettering Cancer Center, New York, New York
  - Vidant Medical Center, Greenville, North Carolina
  - University of Cincinnati (UC) - Cancer Institute, Cincinnati, Ohio
  - The Ohio State University (OSU), Columbus, Ohio
  - Mid Ohio Oncology/Hematology, Inc. dba The Mark H. Zangmeister Center, Columbus, Ohio
  - Williamette Valley Cancer Institute and Research Center, Eugene, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Texas Oncology - Austin Central (Balcones Dr.), Austin, Texas
  - Texas Oncology - DFWW (Bedford), Bedford, Texas
  - Texas Oncology - Fort Worth Cancer Center, Fort Worth, Texas
  - Baylor College of Medicine, Houston, Texas
  - University of Virginia - Emily Couric Cancer Center, Charlottesville, Virginia
  - Virginia Cancer Specialists, PC (Lake Manassas Dr), Gainesville, Virginia
- Australia (7):
  - Cancer Research SA, Adelaide
  - Blacktown Hospital, Blacktown
  - Royal Brisbane and Women's Hospital, Brisbane
  - Epworth HealthCare, East Melbourne
  - Canberra Hospital, Garran
  - Icon Cancer Centre, South Brisbane
  - Wollongong Hospital (Illawarra Shoalhaven Local Health District), Wollongong
- Austria (5):
  - LKH Feldkirch, Feldkirch
  - Medizinische Universitaet Graz, Graz
  - Medizinische Universitaet Innsbruck, Innsbruck
  - Medizinische Universitaet Wien, Vienna
  - Wiener Gesundheitsverbund - Klinik Hietzing, Vienna
- Belgium (6):
  - AZ Klina, Brasschaat
  - Chu Saint-Pierre, Brussels
  - Cliniques Universitaires Saint-Luc, Brussels
  - Clinique CHC MontLégia, Liège
  - AZ Damiaan, Ostend
  - AZ Delta, Roeselare
- Canada (6):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - Juravinski Cancer Centre, Hamilton, Ontario
  - London Health Sciences Centre, London, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - Centre Hospitalier Universite de Sherbrooke (CHUS), Sherbrooke, Quebec
- Czechia (3):
  - Masarykuv onkologicky ustav, Brno
  - Vseobecna fakultni nemocnice v Praze, Prague
  - Fakultni nemocnice Bulovka, Prague
- France (7):
  - Institut de Cancerologie de l'Ouest - site Angers, Angers
  - Centre Leon Berard, Lyon
  - Institut Paoli-Calmettes, Marseille
  - Groupe Hospitalier Diaconesses Croix Saint Simon, Paris
  - Institut de Cancerologie de l'Ouest - site St-Herblain, Saint-Herblain
  - Institut de cancerologie Strasbourg Europe (ICANS), Strasbourg
  - Gustave Roussy, Villejuif
- Germany (8):
  - Charite Universitaetsmedizin Berlin, Berlin
  - Universitaetsklinikum Bonn, Bonn
  - KEM | Evang. Kliniken Essen-Mitte gGmbH, Essen
  - Universitaetsklinikum Heidelberg, Heidelberg
  - Universitaetsklinikum des Saarlandes, Homburg
  - Universitaetsklinikum Schleswig-Holstein Campus Kiel, Kiel
  - Universitaetsmedizin Mannheim, Mannheim
  - Helios Dr. Horst Schmidt Kliniken Wiesbaden, Wiesbaden
- Italy (6):
  - Centro Riferimento Oncologico - Aviano, Aviano
  - Nuovo Ospedale degli Infermi, Ponderano
  - Azienda USL Toscana Centro-Ospedale di Prato Santo Stefano, Prato
  - Fondazione Policlinico Universitario A. Gemelli IRCCS - Universita Cattolica del Sacro Cuore, Rome
  - A.O. Ordine Mauriziano di Torino, Torino
  - Azienda ULSS 2 Marca trevigiana-Ospedale Ca Foncello Treviso, Treviso
- National University Cancer Institute, Singapore, Singapore
- South Korea (8):
  - Keimyung University Dongsan Hospital, Daegu
  - National Cancer Center, Goyang-si
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Samsung Medical Center, Seoul
  - Asan Medical Center, University of Ulsan, Seoul
  - Gangnam Severance Hospital, Yonsei University Health System, Seoul
  - Seoul St. Mary's Hospital, The Catholic University of Korea, Seoul
- Spain (12):
  - Hospital Clinic Barcelona, Barcelona
  - Institut Catala d'Oncologia - L'Hospitalet, Barcelona
  - Institut Catala de Oncologia - Girona, Girona
  - Hospital Universitario Insular de Gran Canaria, Las Palmas de Gran Canaria
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Clinico San Carlos, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - Centro Integral Oncologico Clara Campal, Madrid
  - Hospital Clinico Universitario Virgen de la Arrixaca, Murcia
  - Hospital Clinico Universitario de Valencia, Valencia
  - Hospital Alvaro Cunqueiro, Vigo
- Taiwan (6):
  - Changhua Christian Hospital (CCH), Chang-hua
  - Taichung Veterans General Hospital, Taichung
  - Linkou Chang Gung Memorial Hospital (CGMHLK), Tainan
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
- United Kingdom (5):
  - Cambridge University - Addenbrooke's Hospital, Cambridge
  - University College London Hospital, London
  - Guy's and St Thomas' NHS Foundation Trust, London
  - The Christie NHS Foundation Trust, Manchester
  - Oxford University Hospitals NHS Foundation Trust, Oxford

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Herzog TJ, Hays JL, Barlin JN, Buscema J, Cloven NG, Kong LR, Tyagi NK, Lanneau GS, Long BJ, Marsh RL, Seward SM, Starks DC, Welch S, Moore KN, Konstantinopoulos PA, Gilbert L, Monk BJ, O'Malley DM, Chen X, Dalal R, Coleman RL, Sehouli J. ARTISTRY-7: phase III trial of nemvaleukin alfa plus pembrolizumab vs chemotherapy for platinum-resistant ovarian cancer. Future Oncol. 2023 Jul;19(23):1577-1591. doi: 10.2217/fon-2023-0246. Epub 2023 Jun 19. PMID 37334673

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted globally from 10 Jan 2022 to 08 May 2025.
Pre-assignment Details: Participants with platinum-resistant epithelial ovarian, fallopian tube, or primary peritoneal cancer were enrolled into 1 of 4 arms to receive nemvaleukin alfa (ALKS 4230) either as monotherapy or in combination with pembrolizumab or in investigator's choice chemotherapy. Study was terminated due to business and strategic decision.
Groups:
- Nemvaleukin 6 mcg/kg and Pembrolizumab 200 mg: Participants received Nemvaleukin 6 mcg/kg/day IV infusion over 30 minutes on Days 1 through 5 of 21-day cycles and Pembrolizumab 200 mg IV infusion over 30 minutes on Day 1 of 21-day cycles.
- Pembrolizumab 200 mg: Participants received Pembrolizumab 200 mg IV infusion over 30 minutes on Day 1 of 21-day cycles.
- Nemvaleukin 6 mcg/kg: Participants received Nemvaleukin 6 mcg/kg/day IV infusion over 30 minutes on Days 1 through 5 of 21-day cycles.
- Investigator's Choice Chemotherapy: Investigator's choice chemotherapy includes one of the following: pegylated liposomal doxorubicin (PLD), paclitaxel, topotecan, or gemcitabine. The Investigator pre-selected the Investigator's choice treatment before the randomization of each participant.
  Pegylated Liposomal Doxorubicin (PLD): 40 mg/m^2; Day 1 of 28-day cycles; IV infusion; 1 mg/min (Cycle 1); 60 min infusion (Cycles 2+).
  Paclitaxel: 80 mg/m^2; Days 1, 8, 15, and 22 of 28-day cycles; IV infusion over 60 min.
  Topotecan: 4 mg/m^2; Days 1, 8, and 15 of 28-day cycles; or 1.25 mg/m2, Days 1 through 5 of 21-day cycles; IV infusion over 30 min.
  Gemcitabine: 1,000 mg/m^2; Days 1 and 8 of 21-day cycles; IV infusion over 30 min.
Period: Overall Study
Arm/Group | Nemvaleukin 6 mcg/kg and Pembrolizumab 200 mg | Pembrolizumab 200 mg | Nemvaleukin 6 mcg/kg | Investigator's Choice Chemotherapy
Started | 184 | 27 | 55 | 190
Intent to Treat Population (The intent to treat (ITT) Population will include all randomized participants regardless of the study drug received.) | 184 | 27 | 55 | 190
Safety Set Population (The Safety Population included all randomized participants who received any exposure to nemvaleukin, pembrolizumab, or Investigator's choice chemotherapy.) | 178 | 26 | 53 | 175
Completed | 0 | 0 | 0 | 0
Not Completed | 184 | 27 | 55 | 190
Not completed — Withdrawal by Subject | 21 | 4 | 9 | 26
Not completed — Death | 97 | 14 | 31 | 101
Not completed — Lost to Follow-up | 1 | 2 | 2 | 2
Not completed — Study terminated by sponsor | 65 | 7 | 13 | 61

BASELINE CHARACTERISTICS:
Population: ITT population.
Groups:
- Total: Total of all reporting groups
Arm/Group | Nemvaleukin 6 mcg/kg and Pembrolizumab 200 mg | Pembrolizumab 200 mg | Nemvaleukin 6 mcg/kg | Investigator's Choice Chemotherapy | Total
Number analyzed (Participants) | 184 | 27 | 55 | 190 | 456
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.6 (8.83) | 61.6 (12.97) | 61.5 (9.17) | 61.3 (9.99) | 61.8 (9.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 184 | 27 | 55 | 190 | 456
  Male | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 0 | 2 | 11 | 21
  Not Hispanic or Latino | 165 | 27 | 52 | 175 | 419
  Unknown or Not Reported | 11 | 0 | 1 | 4 | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 0 | 0 | 3
  Asian | 42 | 5 | 3 | 33 | 83
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 1 | 1
  Black or African American | 3 | 0 | 0 | 1 | 4
  White | 113 | 20 | 51 | 142 | 326
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 24 | 1 | 1 | 13 | 39

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: Estimates based on Kaplan-Meier method.
Time Frame: From the first dose of study drug up to 24 months
Population: ITT population.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Nemvaleukin 6 mcg/kg and Pembrolizumab 200 mg | Pembrolizumab 200 mg | Nemvaleukin 6 mcg/kg | Investigator's Choice Chemotherapy
Number analyzed (Participants) | 184 | 27 | 55 | 190
months | 10.1 [7.4 to 12.5] | 10.1 [4.0 to NA] — Higher limit of 95% CI could not be assessed due to the limited number of participants and death events within this reporting group. | 10.7 [8.1 to 13.9] | 9.8 [8.2 to 11.5]

2. Secondary Outcome: Objective Response Rate (ORR) as Assessed by Investigator
Description: Response is based on RECIST v1.1 criteria.
Time Frame: From the first dose of study drug up to 20 months
Population: ITT population.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Nemvaleukin 6 mcg/kg and Pembrolizumab 200 mg | Pembrolizumab 200 mg | Nemvaleukin 6 mcg/kg | Investigator's Choice Chemotherapy
Number analyzed (Participants) | 184 | 27 | 55 | 190
percentage of participants | 9.2 [5.5 to 14.4] | 0.0 [0.0 to 6.5] | 0.0 [00 to 12.8] | 11.1 [7.0 to 16.4]

3. Secondary Outcome: Disease Control Rate (DCR) as Assessed by Investigator
Description: Response is based on RECIST v1.1 criteria.
Time Frame: From the first dose of study drug up to 20 months
Population: ITT population.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Nemvaleukin 6 mcg/kg and Pembrolizumab 200 mg | Pembrolizumab 200 mg | Nemvaleukin 6 mcg/kg | Investigator's Choice Chemotherapy
Number analyzed (Participants) | 184 | 27 | 55 | 190
percentage of participants | 34.2 [27.4 to 41.6] | 25.9 [11.1 to 46.3] | 36.4 [23.8 to 50.4] | 52.1 [44.8 to 59.4]

4. Secondary Outcome: Duration of Response (DOR) as Assessed by Investigator
Description: Response is based on RECIST v1.1 criteria.
Time Frame: From the first dose of study drug up to 20 months
Population: ITT population. Here N refers to number of participants with response and were analyzed for this outcome measure.
Measure: Median (Full Range); unit: months
Arm/Group | Nemvaleukin 6 mcg/kg and Pembrolizumab 200 mg | Pembrolizumab 200 mg | Nemvaleukin 6 mcg/kg | Investigator's Choice Chemotherapy
Number analyzed (Participants) | 17 | 0 | 0 | 21
months | 5.9 [2.1 to 14.7] |  |  | 5.4 [1.4 to 12.6]

5. Secondary Outcome: Time to Response (TTR) as Assessed by Investigator
Description: Response is based on RECIST v1.1 criteria.
Time Frame: From the first dose of study drug up to 20 months
Population: ITT population. Here N refers to number of participants with response and were analyzed for this outcome measure.
Measure: Median (Full Range); unit: months
Arm/Group | Nemvaleukin 6 mcg/kg and Pembrolizumab 200 mg | Pembrolizumab 200 mg | Nemvaleukin 6 mcg/kg | Investigator's Choice Chemotherapy
Number analyzed (Participants) | 17 | 0 | 0 | 21
months | 2.83 [1.4 to 5.7] |  |  | 1.64 [1.3 to 10.9]

6. Secondary Outcome: Percentage of Participants With Cancer Antigen (CA)-125 Response as Defined by the Gynecologic Cancer Inter Group (GCIG)
Description: A Cancer Antigen-125 response is defined as at least a 50% reduction in CA-125 levels from baseline, and the response must be confirmed and maintained for at least 28 days as per the GCIG.
Time Frame: From the first dose of study drug up to 20 months
Population: ITT population.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Nemvaleukin 6 mcg/kg and Pembrolizumab 200 mg | Pembrolizumab 200 mg | Nemvaleukin 6 mcg/kg | Investigator's Choice Chemotherapy
Number analyzed (Participants) | 184 | 27 | 55 | 190
percentage of participants | 4.3 [1.9 to 8.4] | 0.0 [0.0 to 12.8] | 0.0 [0.0 to 6.5] | 13.2 [8.7 to 18.8]

7. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Time Frame: From first dose of study drug up to 90 days after last dose (up to 23 months)
Population: Safety Set population.
Measure: Count of Participants; unit: Participants
Arm/Group | Nemvaleukin 6 mcg/kg and Pembrolizumab 200 mg | Pembrolizumab 200 mg | Nemvaleukin 6 mcg/kg | Investigator's Choice Chemotherapy
Number analyzed (Participants) | 178 | 26 | 53 | 175
Participants | 177 | 23 | 51 | 171

8. Secondary Outcome: Progression-free Survival (PFS) as Assessed by Investigator
Time Frame: From the first dose of study drug up to 20 months
Population: ITT population.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Nemvaleukin 6 mcg/kg and Pembrolizumab 200 mg | Pembrolizumab 200 mg | Nemvaleukin 6 mcg/kg | Investigator's Choice Chemotherapy
Number analyzed (Participants) | 184 | 27 | 55 | 190
months | 1.5 [1.4 to 1.7] | 1.5 [1.4 to 2.4] | 1.5 [1.3 to 2.6] | 2.9 [2.6 to 4.0]

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to 90 days after last dose (up to 23 months)
Description: ITT set.
Arm/Group | Nemvaleukin 6 mcg/kg and Pembrolizumab 200 mg | Pembrolizumab 200 mg | Nemvaleukin 6 mcg/kg | Investigator's Choice Chemotherapy
All-Cause Mortality (participants affected / at risk) | 104/184 | 15/27 | 34/55 | 105/190
Serious Adverse Events (participants affected / at risk) | 74/184 | 8/27 | 17/55 | 51/190
Other Adverse Events (participants affected / at risk) | 177/184 | 23/27 | 51/55 | 171/190
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nemvaleukin 6 mcg/kg and Pembrolizumab 200 mg (N=184) | Pembrolizumab 200 mg (N=27) | Nemvaleukin 6 mcg/kg (N=55) | Investigator's Choice Chemotherapy (N=190)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac tamponade (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myocarditis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pericarditis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 4 (4) | 0 (0) | 1 (1) | 3 (3)
Ascites (Gastrointestinal disorders) | 5 (5) | 1 (1) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Duodenal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Faecaloma (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 3 (3) | 0 (0) | 1 (1) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 6 (6) | 0 (0) | 1 (1) | 4 (4)
Intestinal perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intestinal pseudo-obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intestinal stenosis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Large intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Malignant gastrointestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Melaena (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Rectal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 3 (3) | 1 (1) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 6 (6) | 0 (0) | 0 (0) | 3 (3)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
General physical health deterioration (General disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Localised oedema (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 4 (4) | 0 (0) | 0 (0) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hepatitis (Hepatobiliary disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Cytokine release syndrome (Immune system disorders) | 7 (7) | 0 (0) | 1 (1) | 0 (0)
Bacteraemia (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Biliary tract infection (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Catheter site infection (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diverticulitis (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Empyema (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Enterobacter sepsis (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Erysipeloid (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infection (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Influenza (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Immune system disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Pulmonary sepsis (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyelonephritis (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Salmonella sepsis (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Immune system disorders) | 2 (2) | 1 (1) | 1 (1) | 3 (3)
Septic shock (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Wound infection bacterial (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
C-reactive protein increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Liver function test increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Fasciitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intestinal metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Paraneoplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Memory impairment (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 3 (3) | 1 (1) | 2 (2) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal impairment (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Renal injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0) | 0 (0) | 4 (4)
Malignant pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 3 (3) | 0 (0) | 8 (8)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pulmonary venous thrombosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dermatomyositis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Capillary leak syndrome (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lymphocele (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Subclavian vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vasculitis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vena cava thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nemvaleukin 6 mcg/kg and Pembrolizumab 200 mg (N=184) | Pembrolizumab 200 mg (N=27) | Nemvaleukin 6 mcg/kg (N=55) | Investigator's Choice Chemotherapy (N=190)
Anaemia (Blood and lymphatic system disorders) | 53 (102) | 3 (3) | 15 (31) | 64 (165)
Leukopenia (Blood and lymphatic system disorders) | 7 (23) | 1 (1) | 7 (30) | 10 (38)
Lymphopenia (Blood and lymphatic system disorders) | 27 (60) | 0 (0) | 5 (12) | 3 (3)
Neutropenia (Blood and lymphatic system disorders) | 53 (180) | 0 (0) | 16 (65) | 60 (158)
Thrombocytopenia (Blood and lymphatic system disorders) | 25 (56) | 1 (1) | 8 (16) | 35 (110)
Sinus tachycardia (Cardiac disorders) | 4 (5) | 0 (0) | 5 (6) | 3 (3)
Abdominal distension (Gastrointestinal disorders) | 17 (21) | 0 (0) | 3 (3) | 14 (14)
Abdominal pain (Gastrointestinal disorders) | 35 (40) | 4 (4) | 13 (18) | 26 (28)
Abdominal pain upper (Gastrointestinal disorders) | 10 (13) | 1 (1) | 1 (1) | 9 (11)
Ascites (Gastrointestinal disorders) | 11 (16) | 1 (1) | 6 (11) | 8 (11)
Constipation (Gastrointestinal disorders) | 35 (45) | 2 (2) | 12 (16) | 30 (40)
Diarrhoea (Gastrointestinal disorders) | 41 (55) | 3 (3) | 9 (16) | 33 (52)
Dry mouth (Gastrointestinal disorders) | 8 (8) | 0 (0) | 3 (3) | 1 (1)
Nausea (Gastrointestinal disorders) | 71 (101) | 3 (3) | 20 (36) | 63 (81)
Stomatitis (Gastrointestinal disorders) | 8 (11) | 0 (0) | 1 (1) | 11 (13)
Vomiting (Gastrointestinal disorders) | 45 (69) | 1 (1) | 22 (32) | 28 (37)
Asthenia (General disorders) | 37 (50) | 0 (0) | 15 (31) | 43 (75)
Chills (General disorders) | 61 (162) | 1 (1) | 15 (30) | 2 (2)
Fatigue (General disorders) | 51 (80) | 4 (4) | 13 (15) | 43 (64)
Mucosal inflammation (General disorders) | 3 (3) | 0 (0) | 2 (2) | 11 (18)
Oedema peripheral (General disorders) | 28 (35) | 1 (1) | 6 (6) | 14 (15)
Pyrexia (General disorders) | 81 (193) | 1 (1) | 19 (60) | 13 (14)
Cytokine release syndrome (Immune system disorders) | 37 (176) | 0 (0) | 10 (29) | 0 (0)
COVID-19 (Infections and infestations) | 11 (11) | 0 (0) | 0 (0) | 4 (4)
Urinary tract infection (Infections and infestations) | 13 (15) | 4 (4) | 4 (4) | 10 (13)
Infusion related reaction (Injury, poisoning and procedural complications) | 31 (88) | 0 (0) | 12 (37) | 1 (1)
Alanine aminotransferase increased (Investigations) | 52 (94) | 2 (2) | 20 (53) | 14 (22)
Aspartate aminotransferase increased (Investigations) | 62 (116) | 1 (1) | 21 (56) | 15 (16)
Blood alkaline phosphatase increased (Investigations) | 18 (29) | 2 (2) | 10 (15) | 5 (6)
Blood bilirubin increased (Investigations) | 4 (6) | 0 (0) | 6 (11) | 1 (1)
Blood creatinine increased (Investigations) | 9 (13) | 1 (1) | 3 (6) | 4 (12)
Gamma-glutamyltransferase increased (Investigations) | 14 (30) | 1 (2) | 9 (39) | 5 (5)
White blood cell count decreased (Investigations) | 13 (34) | 0 (0) | 4 (11) | 12 (21)
Decreased appetite (Metabolism and nutrition disorders) | 31 (36) | 0 (0) | 10 (13) | 24 (30)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (3) | 1 (1) | 3 (5) | 3 (5)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 17 (32) | 1 (1) | 6 (14) | 5 (5)
Hypokalaemia (Metabolism and nutrition disorders) | 11 (16) | 1 (1) | 5 (8) | 11 (12)
Hypomagnesaemia (Metabolism and nutrition disorders) | 16 (25) | 2 (4) | 2 (3) | 13 (28)
Hyponatraemia (Metabolism and nutrition disorders) | 7 (13) | 1 (2) | 5 (12) | 6 (6)
Hypophosphataemia (Metabolism and nutrition disorders) | 11 (13) | 0 (0) | 2 (3) | 2 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 15 (19) | 4 (4) | 5 (5) | 9 (12)
Back pain (Musculoskeletal and connective tissue disorders) | 12 (14) | 1 (1) | 4 (4) | 12 (14)
Myalgia (Musculoskeletal and connective tissue disorders) | 19 (22) | 0 (0) | 4 (4) | 10 (10)
Dizziness (Nervous system disorders) | 15 (22) | 1 (1) | 5 (7) | 7 (8)
Headache (Nervous system disorders) | 25 (31) | 1 (1) | 9 (12) | 13 (16)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 19 (24)
Insomnia (Psychiatric disorders) | 7 (7) | 0 (0) | 2 (2) | 12 (13)
Pelvic pain (Reproductive system and breast disorders) | 4 (5) | 0 (0) | 3 (3) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 12 (13) | 2 (2) | 1 (1) | 9 (11)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 27 (40) | 5 (7) | 3 (4) | 21 (29)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 0 (0) | 0 (0) | 9 (10)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 (6) | 1 (1) | 3 (3) | 7 (9)
Alopecia (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 0 (0) | 21 (24)
Pruritus (Skin and subcutaneous tissue disorders) | 15 (18) | 0 (0) | 0 (0) | 7 (9)
Rash (Skin and subcutaneous tissue disorders) | 9 (9) | 1 (1) | 2 (2) | 12 (15)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 9 (20) | 0 (0) | 0 (0) | 4 (4)
Hypertension (Vascular disorders) | 10 (35) | 1 (3) | 3 (3) | 4 (4)
Hypotension (Vascular disorders) | 13 (32) | 1 (1) | 5 (5) | 2 (2)

LIMITATIONS AND CAVEATS:
Study was terminated due to business and strategic decision.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2024-01-31): https://cdn.clinicaltrials.gov/large-docs/60/NCT05092360/Prot_000.pdf
  • Statistical Analysis Plan (2024-08-19): https://cdn.clinicaltrials.gov/large-docs/60/NCT05092360/SAP_001.pdf